CLINICAL TRIAL: NCT02590900
Title: Disposition of Intravenous Paracetamol in Young Women, Including During Pregnancy, in Postpartum or When on Oral Contraceptives
Brief Title: Disposition of Intravenous Paracetamol in Young Women
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: ML6563
Record Dates: First submitted 2015-10-19; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Pain
Keywords: pharmacokinetics; pregnancy; oral contraceptives; oestradiol
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- at delivery: women who underwent cesarean at delivery, and needed iv paracetamol as part of multimodal analgesia. In these cases, paracetamol was administered q6h (2g loading dose, 1g q6h for 24 h), and blood and urine samples were collected to describe paracetamol disposition at delivery.
  Interventions: Drug: intravenous paracetamol (acetaminophen)
- postpartum: a subgroup of 8 women initially included in at delivery, underwent a second PK study 2-3 months postpartum and another PK study about 1 year after delivery. This PK study was based on a single iv paracetamol administration (2 g), and blood and urine samples were collected to describe paracetamol disposition in postpartum
  Interventions: Drug: intravenous paracetamol (acetaminophen)
- healthy female volunteers: a group of 8 young healthy women not on oral contraceptives underwent a single PK study (2 g intravenous paracetamol) and blood and urine samples were collected to described paracetamol disposition in healthy female volunteers, not on oral contraceptives.
  Raw data as published by Gregoire et al (Clin Pharm Ther 2007) were available in 14 young women, all on contraceptives.
  Interventions: Drug: intravenous paracetamol (acetaminophen)

INTERVENTIONS:
Drug: intravenous paracetamol (acetaminophen) — paracetamol disposition in young women, exploring the impact of covariates (pregnancy, postpartum, oral contraceptives) in this population.
  Other Names: Perfusalgan, paracetamol Fresenius,

SUMMARY:
Compared to early postpartum (10-15 weeks) observations, paracetamol clearance was significantly higher (21.1 vs 11.7 l.h-1, + 80 %) at delivery. This higher clearance was due to a disproportional increase in glucuronidation (11.6 vs 4.76 l.h-1, + 144 %), a proportional increase in oxidation clearance (4.95 vs 2.77 l.h-1, 78 %) and primary renal clearance (1.15 vs 0.75 l.h-1, 53 %) [KUlo et al, Int J Obstet Anesth]. This increase in glucuronidation clearance may in part be driven by oestradiol, and may explain within and between individual differences in paracetamol metabolism (e.g. oral contraceptives, follicular vs luteal phase, postpartum, pregnancy, or duration of pregnancy) in young women.

Based on a pooled analysis, investigators aimed to further explore the impact of these covariates on paracetamol metabolism based on plasma and urine collections in women at delivery, in postpartum (early, or late) and healthy volunteers, either or not on oral contraceptives (OC) following intravenous (iv) paracetamol administration.

DETAILED DESCRIPTION:
This study aims to perform a pooled analysis of:

1. Paracetamol PK data recently published in 47 pregnant women. In these cases, iv paracetamol was administered q6h after delivery (caesarean) for 24 h. 8 were recruited a second time for an additional single dose pK study in postpartum (Kulo et al, Br J Clin Pharmacol 2013).
2. The PK data as initially published by Gregoire et al, but limited to female volunteers, all on oral contraceptives (n=14) (Gregoire et al, Clin Pharm Ther 2007)
3. A dataset in 8 young women not on oral contraceptives, iv paracetamol, single dose.

ELIGIBILITY:
Inclusion Criteria:

1. informed consent
2. for patients (pregnant women at delivery), there has to be a clinical indication (post caesarean analgesia, NPO) to administer iv paracetamol.

Exclusion Criteria:

1. intolerance to paracetamol
2. withdrawal of informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pooled analysis of different cohorts of young women who all underwent PK study on paracetamol disposition after iv paracetamol administration.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
paracetamol disposition in young women: total clearance and metabolite specific clearance estimates | 24 h is the maximal time frame of this pharmacokinetic study (PK is the outcome measured
  pooled analysis of plasma and urine paracetamol and paracetamol metabolite data published in literature in young women following iv paracetamol administration. Samples (plasma and urine) will be collected in the 24 h time interval after initiation of intravenous paracetamol administration (time interval of the PK study)

CONTACTS AND LOCATIONS:
Overall Officials: karel allegaert, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

REFERENCES:
- [Result] Beleyn B, Vermeersch S, Kulo A, Smits A, Verbesselt R, de Hoon JN, Van Calsteren K, Allegaert K. Estradiol and weight are covariates of paracetamol clearance in young women. Gynecol Obstet Invest. 2014;77(4):211-6. doi: 10.1159/000358394. Epub 2014 Mar 25. PMID 24686129
- [Result] Kulo A, Peeters MY, Allegaert K, Smits A, de Hoon J, Verbesselt R, Lewi L, van de Velde M, Knibbe CA. Pharmacokinetics of paracetamol and its metabolites in women at delivery and post-partum. Br J Clin Pharmacol. 2013 Mar;75(3):850-60. doi: 10.1111/j.1365-2125.2012.04402.x. PMID 22845052
- [Result] Gregoire N, Hovsepian L, Gualano V, Evene E, Dufour G, Gendron A. Safety and pharmacokinetics of paracetamol following intravenous administration of 5 g during the first 24 h with a 2-g starting dose. Clin Pharmacol Ther. 2007 Mar;81(3):401-5. doi: 10.1038/sj.clpt.6100064. PMID 17339870